CLINICAL TRIAL: NCT05797428
Title: The Effects of Logotherapy on Meaning in Life, Depression, Anxiety and Suicidal Ideation in Adolescents With Mood Disorders
Brief Title: The Effects of Logotherapy in Adolescents With Mood Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Kaoshiung Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202212025RINA
Record Dates: First submitted 2023-03-20; First posted 2023-04-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Mood Disorder of Depressed Type
Keywords: logotherapy; depression; anxiety; suicidal ideation; adolescent
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation | interventions — Logotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Logotherapy (Experimental): 3 months of logotherapy intervention by interviewing with the participant, once every two weeks, about 1-2 hours each time, a total of 6 times of logotherapy.
  Interventions: Other: logotherapy
- Routine psychiatric outpatient treatment (No Intervention): Will not provide any logotherapy. Just routine psychiatric outpatient treatment.

INTERVENTIONS:
Other: logotherapy — The logotherapy is carried out in an individual way in this study. The full-time assistant will give the experimental group 3 months of logotherapy intervention by interviewing with the participant, once every two weeks, about 1-2 hours each time, a total of 6 times of logotherapy to guide the participant to find the meaning of his life and value.The location is mainly in the hospital when the participant has to return for consultation, or at the participant's home.
  Arms: Logotherapy

SUMMARY:
Logotherapy can help people find their meaning in life and help people reduce their suicidal ideation. Suicide was the second leading cause of death for 15-24 year-olds. Logotherapy can increase exploration of meaning in life for adolescents and prevent them from attempting suicide. However, most research only explored the effects of logotherapy on meaning in life and depression in adolescents with mood disorders. There is a lack of research to explore the effects of logotherapy on anxiety and suicidal ideation in adolescents. Therefore, this study will explore the effects of logotherapy on meaning in life, depression, anxiety and suicidal ideation in adolescents with mood disorders. This study will carry on for two years and the sample will be recruited from the adolescents' outpatient clinic of psychiatric department in hospitals. The first and second year of the study will use a single-blind randomized controlled trial approach, the aim is to evaluate the short-term and longitudinal effects of logotherapy meaning in life, depression, anxiety and suicidal ideation in adolescents with mood disorders, the sample will collect 120 adolescents with mood disorders, and will use four instruments for testing the logotherapy intervention. The four instruments are: (1) Purpose in life Test, (2) Beck Depression Inventory II, (3) Beck Anxiety Inventory, (4) Beck Scale for Suicide Ideation. Data will be analyzed using the Statistic Package for the Social Science. The result of this study will be applied to the mental health team in the clinical psychiatric department for taking care of patients, and help adolescents with mood disorders to find their meaning in life, further, to reduce their depression, anxiety and suicidal ideation.

DETAILED DESCRIPTION:
Logotherapy can help people find their meaning in life and help people reduce their suicidal ideation. Suicide was the second leading cause of death for 15-24 year-olds. Logotherapy can increase exploration of meaning in life for adolescents and prevent them from attempting suicide. However, most research only explored the effects of logotherapy on meaning in life and depression in adolescents with mood disorders. There is a lack of research to explore the effects of logotherapy on anxiety and suicidal ideation in adolescents. Therefore, this study will explore the effects of logotherapy on meaning in life, depression, anxiety and suicidal ideation in adolescents with mood disorders. This study will carry on for two years and the sample will be recruited from the adolescents' outpatient clinic of psychiatric department in hospitals. The first and second year of the study will use a single-blind randomized controlled trial approach, the aim is to evaluate the short-term and longitudinal effects of logotherapy meaning in life, depression, anxiety and suicidal ideation in adolescents with mood disorders, the sample will collect 120 adolescents with mood disorders, and will use four instruments for testing the logotherapy intervention. The four instruments are: (1) Purpose in life Test, (2) Beck Depression Inventory II, (3) Beck Anxiety Inventory, (4) Beck Scale for Suicide Ideation. Data will be analyzed using the Statistic Package for the Social Science.

The research process includes:

1. Participant acceptance and signing consent: Referral by doctors from Chang Gung Hospitals and National Taiwan University Hospitals. Full-time research assistants will explain the purpose of the research, the research process, the confidentiality of data processing, and allow the individual to freely decide whether to participate without being forced, obtaining a signed consent form. Those who are under twenty-years-old will also obtain the consent of the legal representative.
2. Pre-test: data collectors blinded single-blind study, the work-students who did not participate in the intervention measures will collect the patient's basic data sheet and four scales.
3. Random assignment: The psychologist (co-host) randomly assigns the cases to the experimental group or the control group, and assigns the groups by means of a computer-generated random assignment table.
4. Intervention: The experimental group received 6 interventions of logotherapy given by a full-time assistant, while the control group received routine outpatient treatment of general adolescent psychiatry.
5. Posttest: Both the experimental group and the control group will collect the same four scales three times by the work-study students.

The result of this study will be applied to the mental health team in the clinical psychiatric department for taking care of patients, and help adolescents with mood disorders to find their meaning in life, further, to reduce their depression, anxiety and suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mood disorders (such as depression, bipolar disorder) diagnosed by a psychiatrist.
* Patient Health Questionnaire-9 items (PHQ-9) score 5-19 points (indicating mild depression to moderate to severe depression)
* Agree to participate in logotherapy
* Able to participate in logotherapy

Exclusion Criteria:

* Patients with severe emotional disorders who cannot participate in logotherapy.
* Those who have severe psychopathological phenomena and cannot judge reality or those who are mentally deficient.
* Those who have serious suicidal ideation or clear suicide plan are not suitable for interview

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Purpose in life Test-1 | pre-test (before intervention)
  There are 20 items in this scale, which are divided into four dimensions: quality of life, value of life, purpose of life, and freedom of life. Each question is scored on a scale of 1-5, and the total score ranges from 20-100, with higher scores representing a higher sense of meaning in life.
Purpose in life Test-2 | post-test 1 (the week after the intervention)
  There are 20 items in this scale, which are divided into four dimensions: quality of life, value of life, purpose of life, and freedom of life. Each question is scored on a scale of 1-5, and the total score ranges from 20-100, with higher scores representing a higher sense of meaning in life.
Purpose in life Test-3 | post-test 2 (three months after the intervention)
  There are 20 items in this scale, which are divided into four dimensions: quality of life, value of life, purpose of life, and freedom of life. Each question is scored on a scale of 1-5, and the total score ranges from 20-100, with higher scores representing a higher sense of meaning in life.
Purpose in life Test-4 | post-test 3 (nine months after the intervention)
  There are 20 items in this scale, which are divided into four dimensions: quality of life, value of life, purpose of life, and freedom of life. Each question is scored on a scale of 1-5, and the total score ranges from 20-100, with higher scores representing a higher sense of meaning in life.
Beck Depression Inventory II-1 | pre-test (before intervention)
  This scale has a total of 21 items. Each item is scored from 0-3 points, and the total score ranges from 0-63 points. The higher the score, the higher the degree of depression.
Beck Depression Inventory II-2 | post-test 1 (the week after the intervention)
  This scale has a total of 21 items. Each item is scored from 0-3 points, and the total score ranges from 0-63 points. The higher the score, the higher the degree of depression.
Beck Depression Inventory II-3 | post-test 2 (three months after the intervention)
  This scale has a total of 21 items. Each item is scored from 0-3 points, and the total score ranges from 0-63 points. The higher the score, the higher the degree of depression.
Beck Depression Inventory II-4 | post-test 3 (nine months after the intervention)
  This scale has a total of 21 items. Each item is scored from 0-3 points, and the total score ranges from 0-63 points. The higher the score, the higher the degree of depression.
Beck Anxiety Inventory-1 | pre-test (before intervention)
  This scale contains 21 items and each item is scored from 0-3 points. The total score ranges from 0-63 points. The higher the score, the higher the degree of anxiety.
Beck Anxiety Inventory-2 | post-test 1 (the week after the intervention)
  This scale contains 21 items and each item is scored from 0-3 points. The total score ranges from 0-63 points. The higher the score, the higher the degree of anxiety.
Beck Anxiety Inventory-3 | post-test 2 (three months after the intervention)
  This scale contains 21 items and each item is scored from 0-3 points. The total score ranges from 0-63 points. The higher the score, the higher the degree of anxiety.
Beck Anxiety Inventory-4 | post-test 3 (nine months after the intervention)
  This scale contains 21 items and each item is scored from 0-3 points. The total score ranges from 0-63 points. The higher the score, the higher the degree of anxiety.
Beck Scale for Suicide Ideation-1 | pre-test (before intervention)
  This scale contains 21 items. The first 19 items mainly measure the severity of the individual's attitudes, behaviors, and plans for suicide in the past week. Each question is calculated on a scale of 0-2, and the total score ranges from 0-38, with higher scores indicating stronger suicidal ideation. The last two questions, which are not counted, ask about the number of previous suicide attempts and the severity of the intention of the last suicide attempt.
Beck Scale for Suicide Ideation-2 | post-test 1 (the week after the intervention)
  This scale contains 21 items. The first 19 items mainly measure the severity of the individual's attitudes, behaviors, and plans for suicide in the past week. Each question is calculated on a scale of 0-2, and the total score ranges from 0-38, with higher scores indicating stronger suicidal ideation. The last two questions, which are not counted, ask about the number of previous suicide attempts and the severity of the intention of the last suicide attempt.
Beck Scale for Suicide Ideation-3 | post-test 2 (three months after the intervention)
  This scale contains 21 items. The first 19 items mainly measure the severity of the individual's attitudes, behaviors, and plans for suicide in the past week. Each question is calculated on a scale of 0-2, and the total score ranges from 0-38, with higher scores indicating stronger suicidal ideation. The last two questions, which are not counted, ask about the number of previous suicide attempts and the severity of the intention of the last suicide attempt.
Beck Scale for Suicide Ideation-4 | post-test 3 (nine months after the intervention)
  This scale contains 21 items. The first 19 items mainly measure the severity of the individual's attitudes, behaviors, and plans for suicide in the past week. Each question is calculated on a scale of 0-2, and the total score ranges from 0-38, with higher scores indicating stronger suicidal ideation. The last two questions, which are not counted, ask about the number of previous suicide attempts and the severity of the intention of the last suicide attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Fan-Ko Sun, PhD, Study Chair — Second Degree Bachelor of Science in nursing, National Taiwan University
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Niaosong District, Taiwan

IPD SHARING:
Plan to Share IPD: No